CLINICAL TRIAL: NCT02198664
Title: Oral Desensitization to Peanut in Peanut-Allergic Children and Adults Using Characterized Peanut Allergen (CPNA) Peanut Oral Immunotherapy (OIT) Safety Follow-On Study
Brief Title: Oral Desensitization to Peanut in Peanut Allergic Children and Adults Using CPNA Peanut OIT Safety Follow-On Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aimmune Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARC002
Record Dates: First submitted 2014-07-22; First posted 2014-07-24 (Estimated); Results first posted 2021-11-09 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Peanut Allergy
Keywords: Characterized Peanut Allergen; Peanut; OIT; Oral Desensitization; Peanut Allergen; Peanut-Allergic Children; Children; Peanut-Allergic Adults
MeSH Terms: conditions — Peanut Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ARC001 placebo group (Experimental): Subjects who received placebo in study ARC001.
  Interventions: Biological: AR101 - Peanut protein capsule
- ARC001 AR101 group (Experimental): Subjects who received AR101 and tolerated up to 300 mg peanut protein (443 mg cumulative) in the DBPCFC at the end of study ARC001.
  Interventions: Biological: AR101 - Peanut protein capsule

INTERVENTIONS:
Biological: AR101 - Peanut protein capsule — Study product provided as peanut protein in pull-apart capsules at 5 dosage strengths (0.5, 1, 10, 100, and 475 mg) or sachets at 2 dosage strengths (300 and 1000 mg)

SUMMARY:
This is a multi-center, open-label, follow-on study to gather additional information on the safety and tolerability of oral desensitization with CPNA in the subjects who participated in ARC001.

DETAILED DESCRIPTION:
This phase 2, open-label, follow-on, multicenter study was designed to gather additional information on the safety, tolerability, and efficacy of oral desensitization with AR101 in subjects who participated in study ARC001 (NCT01987817) as follows:

* Group 1 (ARC001 placebo): Subjects who received placebo in study ARC001
* Group 2 (ARC001 AR101): Subjects who received AR101 and tolerated up to 300 mg peanut protein (443 mg cumulative) in the DBPCFC at the end of study ARC001

All subjects will receive daily oral dosing of peanut OIT (oral immunotherapy) in the form of Characterized Peanut Allergen (CPNA).

Study Duration - 12-90 weeks before reaching the Extended Maintenance Phase. All Subjects may continue Extended Maintenance Phase until CPNA becomes commercially available or the study is terminated.

ELIGIBILITY:
Key Inclusion Criteria:

* Completion of ARC001 study
* No change in the status of any longitudinally applicable ARC001 inclusion criteria

Key Exclusion Criteria:

* Early termination from ARC001
* Failure to tolerate 300 mg of peanut protein in the ARC001 exit food challenge
* A lapse in dosing of more than 10 days from completion of ARC001
* Change in the status of any longitudinally applicable ARC001 exclusion criteria

Ages: 4 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 47 (Actual)
Dates: Start 2014-08-27 (Actual); Primary Completion 2018-01-04 (Actual); Study Completion 2018-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Director of Regulatory Affairs, Study Director — Aimmune Therapeutics
Locations (8):
- United States (8):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - UC San Diego, San Diego, California
  - Boston Children's Hospital, Boston, Massachusetts
  - Mount Sinai Medical Center, New York, New York
  - University of North Carolina Chapel HIll, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Medical Center Dallas, Dallas, Texas

REFERENCES:
- [Derived] Nilsson C, Scurlock AM, Dellon ES, Brostoff JM, Pham T, Ryan R, Brown KR, Adelman DC, Aceves SS. Onset of eosinophilic esophagitis during a clinical trial program of oral immunotherapy for peanut allergy. J Allergy Clin Immunol Pract. 2021 Dec;9(12):4496-4501. doi: 10.1016/j.jaip.2021.07.048. Epub 2021 Aug 11. No abstract available. PMID 34389504

RESULTS

PARTICIPANT FLOW:
Groups:
- ARC001 Placebo Group: Subjects who received placebo in study ARC001.
  AR101 - Peanut protein provided in capsules: Study product provided as peanut protein in pull-apart capsules at 5 dosage strengths (0.5, 1, 10, 100, and 475 mg) or sachets at 2 dosage strengths (300 and 1000 mg)
- ARC001 AR101 Group: Subjects who received AR101 and tolerated up to 300 mg peanut protein (443 mg cumulative) in the DBPCFC at the end of study ARC001.
  AR101 - Peanut protein provided in capsules: Study product provided as peanut protein in pull-apart capsules at 5 dosage strengths (0.5, 1, 10, 100, and 475 mg) or sachets at 2 dosage strengths (300 and 1000 mg)
Period: Overall Study
Arm/Group | ARC001 Placebo Group | ARC001 AR101 Group
Started | 26 | 21
Completed | 10 | 13
Not Completed | 16 | 8
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 11 | 8
Not completed — Failure to tolerate | 2 | 0
Not completed — Not stated | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ARC001 Placebo Group | ARC001 AR101 Group | Total
Number analyzed (Participants) | 26 | 21 | 47
Age, Continuous [Median (Full Range); unit: years] | 8.5 [5.0 to 14.0] | 8.0 [4.0 to 21.0] | 8.0 [4.0 to 21.0]
Age, Customized [Count of Participants; unit: Participants]
  4-17 years | 26 | 20 | 46
  18-26 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 17
  Male | 16 | 14 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 26 | 21 | 47
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 20 | 18 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Adverse Events and Dosing Symptoms Occurring With Peanut OIT Over a Protracted Treatment Period Comprising at Least 18 Months
Description: TEAEs are any event starting during or after the active treatment period. If a subject has multiple occurrences of TEAEs, the subject is presented once in the respective subject count (n).
Time Frame: Up to 90 weeks
Population: The Safety Population (those who received any amount of AR101)
Measure: Count of Participants; unit: Participants
Arm/Group | ARC001 Placebo Group | ARC001 AR101 Group
Number analyzed (Participants) | 26 | 21
Participants
  Any TEAE | 26 | 21
  Any Grade 3 or Higher TEAE | 1 | 1
  Any TEAE Related to Study Treatment | 25 | 15
  Any TEAE Leading to Study Treatment Temporarily Withdrawn | 12 | 15
  Any TEAE Event Leading to Study Treatment Permanently Withdrawn | 4 | 0
  Any Treatment-Related Hypersensitivity Adverse Event | 5 | 4
  Any serious TEAE | 0 | 1
  Any Serious TEAE leading to Death | 0 | 0

2. Secondary Outcome: The Proportion of Subjects Who Tolerated at Least 300 mg (443 mg) and 600 mg (1043 mg Cumulative) Peanut Protein With no More Than Mild Symptoms During the Up-dosing DBPCFC
Time Frame: Up to 36 weeks
Population: The Safety Population (those who received any amount of AR101). Only results for the "ARC001 AR101 Group" is reported as only subjects in this group had Up-dosing DBPCFC in ARC002 study.
Measure: Count of Participants; unit: Participants
Arm/Group | ARC001 Placebo Group
Number analyzed (Participants) | 26
Participants
  Up-dosing DBPCFC: Responder at 300 mg | 20
  Up-dosing DBPCFC: Responder at 600 mg | 19

3. Secondary Outcome: The Proportion of Subjects Who Tolerated at Least 300 mg (443 mg), 600 mg (1043 mg Cumulative), and 1000 mg Peanut Protein (2043 mg Cumulative) With no More Than Mild Symptoms During the Maintenance DBPCFC.
Time Frame: Up to 60 weeks.
Population: The Safety Population (those who received any amount of AR101). Multiple food challenge dose levels were given at each DBPCFC, so results at 300 mg and 600 mg for Maintenance DBPCFC are not expected to match those for Up-dosing DBPCFC.
Measure: Count of Participants; unit: Participants
Arm/Group | ARC001 Placebo Group | ARC001 AR101 Group
Number analyzed (Participants) | 26 | 21
Participants
  Maintenance DBPCFC: Responder at 300 mg | 20 | 20
  Maintenance DBPCC: Responder at 600 mg | 20 | 18
  Maintenance DBPCC: Responder at 1000 mg | 17 | 14

4. Secondary Outcome: Change From Baseline in the Single Highest Tolerated Dose of Peanut Protein
Description: The single highest tolerated dose of peanut protein with no more than mild symptoms during the up-dosing DBPCFC and the change from baseline was evaluated for the ARC001 placebo completer population. The single highest tolerated dose of peanut protein with no more than mild symptoms during the maintenance DBPCFC and the change from up-dosing DBPCFC was evaluated for each group (ARC001 AR101 and ARC001 placebo) and overall for the food challenge completer population.
Time Frame: Up to 60 weeks (Up to 36 weeks for up-dosing; up to 24 weeks for maintenance)
Population: Only includes food challenge completer population
Measure: Geometric Mean (Standard Deviation); unit: mg
Arm/Group | ARC001 Placebo Group | ARC001 AR101 Group
Number analyzed (Participants) | 26 | 21
mg
  AR101 baseline (mg) [2] | 38.90 (4.37) | NA (NA) — 1. Baseline values for ARC001 AR101 group were already summarized in ARC001 and were not re-summarized in ARC002 2. The single highest tolerated dose from the ARC001 exit DBPCFC was defined as the AR101 baseline for subjects in the ARC001 placebo group.
  Up-dosing DBPCFC: number analyzed (Participants) | 21 | 21
  Up-dosing DBPCFC | 501.2 (1.55) | 524.8 (1.32)
  Maintenance DBPCFC: number analyzed (Participants) | 20 | 20
  Maintenance DBPCFC | 776.2 (1.41) | 758.6 (1.55)

5. Secondary Outcome: Number of Participants Who Tolerated Maximum Dose of Peanut Protein With no More Than Mild Symptoms Maximum Dose of Peanut Protein Tolerated
Description: The maximum dose of peanut protein tolerated with no more than mild symptoms during the up-dosing and maintenance DBPCFCs
Time Frame: Up to 60 weeks (Up to 36 weeks for up-dosing; up to 24 weeks for maintenance)
Population: Only includes food challenge completer population
Measure: Count of Participants; unit: Participants
Arm/Group | ARC001 Placebo Group | ARC001 AR101 Group
Number analyzed (Participants) | 26 | 21
Participants
  Up-dosing DBPCFC: number analyzed (Participants) | 21 | 21
  Up-dosing DBPCFC: 100 mg | 1 | 0
  Up-dosing DBPCFC: 300 mg | 3 | 4
  Up-dosing DBPCFC: 600 mg | 17 | 17
  Up-dosing DBPCFC: 1000 mg | NA — Not administer 1000 mg dose at Up-dosing DBPCFC. | NA — Not administer 1000 mg dose at Up-dosing DBPCFC.
  Maintenance DBPCFC: number analyzed (Participants) | 20 | 20
  Maintenance DBPCFC: 100 mg | 0 | 0
  Maintenance DBPCFC: 300 mg | 1 | 3
  Maintenance DBPCFC: 600 mg | 8 | 4
  Maintenance DBPCFC: 1000 mg | 11 | 13

6. Secondary Outcome: Change in Peanut-specific IgE From Baseline and Up-dosing to Extended Maintenance
Time Frame: Baseline, Up-dosing (up to 36 weeks), Extended Maintenance (up to 90 weeks)
Population: The Safety Population (those who received any amount of AR101)
Measure: Geometric Mean (Standard Deviation); unit: kU/L
Arm/Group | ARC001 Placebo Group | ARC001 AR101 Group
Number analyzed (Participants) | 26 | 21
kU/L
  Baseline: Peanut-specific IgE | 56.826 (2.8864) | NA (NA) — [1] Baseline values for ARC001 AR101 group were already summarized in ARC001 and were not re-summarized in ARC002
  Up-dosing: Peanut-specific IgE | 59.145 (2.9154) | 29.964 (4.4817)
  Extended maintenance: Peanut-specific IgE | 14.880 (6.7531) | 10.381 (4.0149)
  Change from baseline: Peanut-specific IgE | 0.387 (2.2479) | NA (NA) — [1] Baseline values for ARC001 AR101 group were already summarized in ARC001 and were not re-summarized in ARC002
  Change from up-dosing: Peanut-specific IgE | 0.364 (2.8292) | 0.228 (2.0544)

7. Secondary Outcome: Change in Peanut-specific IgG4 From Baseline and Up-dosing to Extended Maintenance
Time Frame: Baseline, Up-dosing (up to 36 weeks), Extended Maintenance (up to 90 weeks)
Population: The Safety Population (those who received any amount of AR101)
Measure: Geometric Mean (Standard Deviation); unit: μg/mL
Arm/Group | ARC001 Placebo Group | ARC001 AR101 Group
Number analyzed (Participants) | 26 | 21
μg/mL
  Baseline: Peanut-specific IgG4 | 0.538 (2.4351) | NA (NA) — Baseline values for ARC001 AR101 group were already summarized in ARC001 and were not re-summarized in ARC002
  Up-dosing: Peanut-specific IgG4 | 3.004 (3.8962) | 4.096 (3.9749)
  Extended maintenance: Peanut-specific IgG4 | 5.755 (3.6328) | 12.429 (2.8292)
  Change from baseline: Peanut-specific IgG4 | 12.429 (2.2705) | NA (NA) — Baseline values for ARC001 AR101 group were already summarized in ARC001 and were not re-summarized in ARC002
  Change from up-dosing: Peanut-specific IgG4 | 1.682 (3.1268) | 2.746 (3.4556)

8. Secondary Outcome: Change in Skin Prick Test (SPT) Mean Peanut Wheal Diameter and Peanut Erythema/Flare From Baseline and Up-dosing to Extended Maintenance
Time Frame: Baseline, Up-dosing (up to 36 weeks), Extended Maintenance (up to 90 weeks)
Population: The Safety Population (those who received any amount of AR101)
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | ARC001 Placebo Group | ARC001 AR101 Group
Number analyzed (Participants) | 26 | 21
millimeter
  Peanut wheal diameter; baseline | 11.8 (6.29) | NA (NA) — Baseline values for ARC001 AR101 group were already summarized in ARC001 and were not re-summarized in ARC002
  Peanut wheal diameter; up-dosing | 8.6 (4.62) | 6.6 (3.04)
  Peanut wheal diameter; extended maintenance | 9.0 (5.77) | 5.1 (3.40)
  Change from baseline: Peanut wheal diameter | -1.5 (6.52) | NA (NA) — Baseline values for ARC001 AR101 group were already summarized in ARC001 and were not re-summarized in ARC002
  Change from up-dosing: Peanut wheal diameter | -0.8 (4.72) | -0.7 (2.98)
  Peanut erythema/flare; baseline | 37.6 (17.69) | NA (NA) — Baseline values for ARC001 AR101 group were already summarized in ARC001 and were not re-summarized in ARC002
  Peanut erythema/flare; up-dosing | 26.8 (12.05) | 21.8 (8.76)
  Peanut erythema/flare; extended maintenance | 28.2 (19.73) | 14.7 (11.62)
  Change from baseline: peanut erythema/flare | -8.7 (15.35) | NA (NA) — Baseline values for ARC001 AR101 group were already summarized in ARC001 and were not re-summarized in ARC002
  Change from up-dosing: peanut erythema/flare | -1.8 (11.55) | -5.4 (9.79)

9. Secondary Outcome: Number of Participants With Maximum Symptom Severity at Each Challenge Dose of Peanut Protein in All Subjects During Up-Dosing DBPCFC
Description: Maximum severity of symptoms that occurred at each challenge dose of peanut protein for all subjects during up-dosing DBPCFC
Time Frame: Up to 36 weeks for up-dosing
Population: Only subjects who completed the food challenge at each challenge dose during the Up-dosing DBPCFC were analyzed
Measure: Count of Participants; unit: Participants
Groups:
- ARC001 Placebo Group: Subjects who received placebo in study ARC001.
  AR101 - Peanut protein provided in capsules: Study product provided as peanut protein in pull-apart capsules at 5 dosage strengths (0.5, 1, 10, 100, and 475 mg) or sachets at 2 dosage strengths (300 and 1000 mg
Arm/Group | ARC001 Placebo Group | ARC001 AR101 Group
Number analyzed (Participants) | 21 | 21
Participants
  3 mg: None | 11 | 18
  3 mg: Mild | 0 | 3
  3 mg: Moderate | 0 | 0
  3 mg: Severe | 0 | 0
  3 mg: Missing | 10 | 0
  10 mg: None | 10 | 21
  10 mg: Mild | 1 | 0
  10 mg: Moderate | 0 | 0
  10 mg: Severe | 0 | 0
  10 mg: Missing | 10 | 0
  30 mg: None | 10 | 20
  30 mg: Mild | 2 | 1
  30 mg: Moderate | 0 | 0
  30 mg: Severe | 0 | 0
  30 mg: Missing | 9 | 0
  100 mg: None | 11 | 18
  100 mg: Mild | 1 | 3
  100 mg: Moderate | 0 | 0
  100 mg: Severe | 0 | 0
  100 mg: Missing | 9 | 0
  300 mg: None | 7 | 20
  300 mg: Mild | 4 | 1
  300 mg: Moderate | 0 | 0
  300 mg: Severe | 0 | 0
  300 mg: Missing | 10 | 0
  600 mg: None | 6 | 12
  600 mg: Mild | 6 | 5
  600 mg: Moderate | 0 | 4
  600 mg: Severe | 0 | 0
  600 mg: Missing | 9 | 0

10. Secondary Outcome: Number of Participants With Maximum Symptom Severity at Each Challenge Dose of Peanut Protein in All Subjects During Maintenance DBPCFC
Description: Maximum severity of symptoms that occurred at each challenge dose of peanut protein for all subjects during maintenance DBPCFC
Time Frame: Up to 60 weeks (Up to 36 weeks for up-dosing; up to 24 weeks for maintenance)
Population: Only subjects who completed the food challenge at each challenge dose during the Maintenance DBPCFC were analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | ARC001 Placebo Group | ARC001 AR101 Group
Number analyzed (Participants) | 20 | 20
Participants
  3 mg: None | 7 | 9
  3 mg: Mild | 0 | 1
  3 mg: Moderate | 0 | 0
  3 mg: Severe | 0 | 0
  3 mg: Missing | 13 | 10
  10 mg: None | 6 | 9
  10 mg: Mild | 0 | 0
  10 mg: Moderate | 0 | 0
  10 mg: Severe | 0 | 0
  10 mg: Missing | 14 | 11
  30 mg: None | 6 | 9
  30 mg: Mild | 0 | 1
  30 mg: Moderate | 0 | 0
  30 mg: Severe | 0 | 0
  30 mg: Missing | 14 | 10
  100 mg: None | 6 | 9
  100 mg: Mild | 1 | 0
  100 mg: Moderate | 0 | 0
  100 mg: Severe | 0 | 0
  100 mg: Missing | 13 | 11
  300 mg: None | 6 | 8
  300 mg: Mild | 0 | 1
  300 mg: Moderate | 0 | 0
  300 mg: Severe | 0 | 0
  300 mg: Missing | 14 | 11
  600 mg: None | 7 | 7
  600 mg: Mild | 2 | 3
  600 mg: Moderate | 0 | 1
  600 mg: Severe | 0 | 0
  600 mg: Missing | 11 | 9
  1000 mg: None | 5 | 7
  1000 mg: Mild | 7 | 4
  1000 mg: Moderate | 2 | 2
  1000 mg: Severe | 0 | 1
  1000 mg: Missing | 6 | 6

11. Secondary Outcome: Change in Physician Global Assessment, Disease Activity as Measured on a 100 mm Visual Analogue Scale (VAS) From Baseline and Up-dosing to Extended Maintenance.
Description: A 100-mm Visual Analog Scale (VAS) was used by the investigators for the Physician Global Assessment of disease activity as a marker for safety. The investigator was to assign a single integrated overall disease activity score ranging from 0 to 100 mm. Zero indicated no disease activity and 100 indicated very severe disease activity.
Time Frame: Baseline, Up-dosing (up to 36 weeks), Extended Maintenance (up to 90 weeks)
Population: The Safety Population (those who received any amount of AR101)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ARC001 Placebo Group | ARC001 AR101 Group
Number analyzed (Participants) | 26 | 21
score on a scale
  Baseline | 36.4 (24.31) | NA (NA) — [1] Baseline values for ARC001 AR101 group were already summarized in ARC001 and were not re-summarized in ARC002
  Up-dosing | 34.9 (21.42) | 25.6 (17.78)
  Extended maintenance | 27.5 (25.03) | 20.1 (12.61)
  Change from baseline | -26.30 (34.50) | NA (NA) — [1] Baseline values for ARC001 AR101 group were already summarized in ARC001 and were not re-summarized in ARC002
  Change from up-dosing | -20.00 (38.87) | -15.5 (20.56)

ADVERSE EVENTS:
Time Frame: 90 weeks
Description: A multi-page adverse event form was used allowing all adverse events to be submitted through a single reporting mechanism. Study investigators will provide the Coordinating Center with data of all SAEs as defined per the protocol on an ongoing basis, within 24 h of site awareness of the event. The sponsor's Medical Monitor will review each SAE report and will determine whether the SAE must be reported to FDA on an expedited basis.
Arm/Group | ARC001 Placebo Group | ARC001 AR101 Group
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/26 | 1/21
Other Adverse Events (participants affected / at risk) | 26/26 | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ARC001 Placebo Group (N=26) | ARC001 AR101 Group (N=21)
Anaphylactic reaction (Immune system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ARC001 Placebo Group (N=26) | ARC001 AR101 Group (N=21)
Abdominal pain (Gastrointestinal disorders) | 15 | 9
Vomiting (Gastrointestinal disorders) | 15 | 8
Abdominal pain upper (Gastrointestinal disorders) | 7 | 7
Nausea (Gastrointestinal disorders) | 7 | 6
Oral pruritus (Gastrointestinal disorders) | 6 | 2
Abdominal discomfort (Gastrointestinal disorders) | 3 | 3
Diarrhoea (Gastrointestinal disorders) | 3 | 3
Lip swelling (Gastrointestinal disorders) | 4 | 2
Dyspepsia (Gastrointestinal disorders) | 3 | 1
Constipation (Gastrointestinal disorders) | 2 | 1
Gastritis (Gastrointestinal disorders) | 2 | 1
Lip pruritus (Gastrointestinal disorders) | 1 | 2
Pharyngitis streptococcal (Infections and infestations) | 10 | 5
Upper respiratory tract infection (Infections and infestations) | 7 | 8
Gastroenteritis viral (Infections and infestations) | 4 | 5
Viral infection (Infections and infestations) | 5 | 4
Gastroenteritis (Infections and infestations) | 3 | 5
Nasopharyngitis (Infections and infestations) | 4 | 4
Otitis media (Infections and infestations) | 3 | 2
Ear infection (Infections and infestations) | 2 | 2
Influenza (Infections and infestations) | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 9 | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Sneezing (Respiratory, thoracic and mediastinal disorders) | 8 | 3
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 7 | 2
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 7 | 5
Rash (Skin and subcutaneous tissue disorders) | 5 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 4
Eczema (Skin and subcutaneous tissue disorders) | 1 | 3
Erythema (Skin and subcutaneous tissue disorders) | 2 | 1
Pyrexia (General disorders) | 7 | 6
Chest discomfort (General disorders) | 1 | 2
Malaise (General disorders) | 1 | 2
Hypersensitivity (Immune system disorders) | 6 | 7
Anaphylactic reaction (Immune system disorders) | 4 | 2
Seasonal allergy (Immune system disorders) | 1 | 3
Food allergy (Immune system disorders) | 0 | 3
Headache (Nervous system disorders) | 6 | 8
Arthropod bite (Injury, poisoning and procedural complications) | 3 | 1
Joint injury (Injury, poisoning and procedural complications) | 2 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 1
Eye pruritus (Eye disorders) | 1 | 2
Ear pruritus (Ear and labyrinth disorders) | 3 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 3 | 0
Flushing (Vascular disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
* Institutions cannot publish until the multi-center sponsor publication is published
* Or, institutions cannot publish until 18 months after study completion
* And Sponsor review of any publications is required prior to any institution publications according to contractual agreements

DOCUMENTS (2):
  • Study Protocol (2017-08-15): https://cdn.clinicaltrials.gov/large-docs/64/NCT02198664/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-02): https://cdn.clinicaltrials.gov/large-docs/64/NCT02198664/SAP_001.pdf